CLINICAL TRIAL: NCT04301830
Title: Postoperative Changes in Optic Nerve Sheath Diameter in Patients Undergoing Spinal Anesthesia for Cesarean Delivery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Other Study IDs: 20200306
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal anesthesia: Patients undergoing cesarean section under spinal anesthesia

SUMMARY:
This is observational study. The investigator will measure optic nerve sheath diameter by ultrasound on the eye after cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients has ophthalmic diseases
* Patients has previous history of ophthalmic surgery.
* Patients has neurological disorders.
* Patients has history of head surgery.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cesarean section under spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change optic nerve sheath diameter | 0,1,6,24 and 48 hours
  Change in Optic nerve sheathe diameter from baseline, 1,,6,24 and 48 hours after completion of surgery

REFERENCES:
- [Background] Watanabe A, Horikoshi T, Uchida M, Ishigame K, Kinouchi H. Decreased diameter of the optic nerve sheath associated with CSF hypovolemia. AJNR Am J Neuroradiol. 2008 May;29(5):863-4. doi: 10.3174/ajnr.A1027. Epub 2008 Feb 29. PMID 18310231
- [Background] Bauerle J, Gizewski ER, Stockhausen Kv, Rosengarten B, Berghoff M, Grams AE, Kaps M, Nedelmann M. Sonographic assessment of the optic nerve sheath and transorbital monitoring of treatment effects in a patient with spontaneous intracranial hypotension: case report. J Neuroimaging. 2013 Apr;23(2):237-9. doi: 10.1111/j.1552-6569.2011.00640.x. Epub 2011 Sep 1. PMID 21883624